CLINICAL TRIAL: NCT00948857
Title: A Randomized Double Blinded Trail of DHEA Supplementation for Treatment of Couples With Premature Ovarian Failure (POF).
Brief Title: Dehydroepiandrosterone (DHEA) Treatment and Premature Ovarian Failure (POF)
Acronym: DHEAFert2
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of recruitment.
Sponsor: David H. Barad (Other)
Responsible Party: Sponsor-Investigator, David H. Barad, Director of Clinical Research, Center for Human Reproduction
Organization: Center for Human Reproduction (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 092508-01
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Premature Ovarian Failure
Keywords: DHEA; POF; Pregnancy; Ovarian Failure; Otherwise Unexplained infertility; Ovarian aging
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DHEA active treatment (Experimental): Dehydroepiandrosterone 25 mg tid po
  Interventions: Dietary Supplement: Dehydroepiandrosterone
- DHEA Placebo (Placebo Comparator): Blinded placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Dehydroepiandrosterone — 25 mg PO TID
  Other Names: DHEA
  Arms: DHEA active treatment
Dietary Supplement: Placebo — Blinded placebo
  Arms: DHEA Placebo

SUMMARY:
The experimental focus of this project is on the interaction of DHEA treatment on pregnancy in women with open tubes, fertile male partners and evidence of premature ovarian failure.

DETAILED DESCRIPTION:
Recruitment:

* New patients presenting for Donor egg cycles
* Possible print, magazine or Radio advertisement

Experimental plan:

1. Informed consent
2. Baseline studies

   * Antral follicle counts
   * Serum FSH, LH, E2, Prog, DHEA, DHEAS, testosterone, AMH, Fragile X
3. Randomization

   * Group A: DHEA (25 mg three times per day)
   * Group B: Placebo
4. Monitoring during treatment

   * All participants will have:
   * USG for follicle measurement
   * Repeat serum, FSH, E2, DHEA, DHEAS, testosterone, AMH monthly during treatment.
   * Physical examination
   * Completion of study questionnaire regarding possible androgen effects of treatment
5. Analysis plan:

   * Primary Outcome
   * Pregnancy
   * Pregnancy rates will be compared using logistic regression with age and pre-treatment AMH as covariates.
   * Secondary Outcomes
   * Endocrine Factors
   * Androgen side effects
   * Primary analysis. We will perform a factorial ANOVA for the two pretreatment factors DHEA and Placebo. Baseline AMH and age as main covariates
   * Secondary analysis.
   * Examine rate of change of estradiol and other endocrine response over the four cycles of treatment
   * Compare antral follicle counts across cycles between groups
   * Compare possible androgen related effects
   * Power considerations:
   * Power assumptions: alpha 0.05; 80% power

Spontaneous Pregnancy rate for POF is less than 1% per 3 months Intervention will improve pregnancy rate to 10% per 3 months. Patients will be treated for 3 cycles. Require 100 patients to complete treatment in each group. Allow for 20% dropout will need 120 patients randomized to each group

* Randomization:

Randomization will be by permuted blocks in order to maintain an even distribution among the groups (because of the small numbers of participants)

* Human subjects issues
* Potential risks associated with DHEA use
* Potential risk of delay of treatment for 3 months and possible natural continued loss of fertility
* Informed consent issues

ELIGIBILITY:
Inclusion Criteria:

* >= 1 year of infertility
* >21 and <40 years old
* Normal HSG
* Normal Semen analysis (Count >= 20 million/ motility > 50%/ Kruger morph > 14%.
* Absent menses
* Willingness to sign informed consent for study randomization
* Willingness to participate in 3 months of treatment.

Exclusion Criteria:

* Abnormal semen analysis
* Abnormal HSG
* Medical condition that would contraindicate pregnancy, ovulation induction or general anesthesia
* Family history of significant genetic disease, or factor V leiden thrombophilia
* Inability to present for monitoring visits
* Inability to follow medication instruction
* Desire to undergo other fertility treatments before completing three months of this trial

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Barad, MD, MS, Principal Investigator — Center for Human Reproduction; Norbert Gleicher, MD, Study Chair — Center for Human Reproduction
Locations (1):
- Center for Human Reproduction, New York, New York, United States

REFERENCES:
- See also: Center for Human Reproduction — http://www.centerforhumanreprod.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Dehydroepiandrosterone 25 mg Tid po: Dehydroepiandrosterone 25 mg tid po
- Blinded Placebo: Blinded placebo
Period: Overall Study
Arm/Group | Dehydroepiandrosterone 25 mg Tid po | Blinded Placebo
Started | 3 | 2
Completed | 2 (3 completed and 1 dropped out.) | 2
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dehydroepiandrosterone 25 mg Tid po | Blinded Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38 (3) | 38 (3) | 38 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Live Birth
Time Frame: 24 months
Reporting Status: Not Posted

2. Secondary Outcome: Endocrine Effects
Time Frame: 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Androgen Side Effects
Time Frame: 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Clinical Pregnancy
Time Frame: 12 months
Reporting Status: Not Posted

5. Primary Outcome: Live Birth
Description: Live Birth outcome compared between DHEA active treatment and Placebo
Time Frame: 9 months
Population: This study was closed for futility because of difficulty finding patients willing to undergo randomization.
Measure: Number; unit: participants
Groups:
- DHEA: Dehydroepiandrosterone 25 mg tid po
Arm/Group | DHEA | Placebo
Number analyzed (Participants) | 3 | 2
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dehydroepiandrosterone 25 mg Tid po | Blinded Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Termination due to lack of consenting participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes